CLINICAL TRIAL: NCT06967493
Title: "Amazonian Dance for Parkinson": a Protocol Study for a Randomized Clinical Trial on Motor and Non-motor Symptoms of People With Parkinson's.
Brief Title: Effects of Amazonian Dance on Motor and Non-motor Symptoms of People With Parkinson's: Study Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Aline Nogueira Haas, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 75675023.9.0000.5327
Record Dates: First submitted 2025-04-18; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: Dance; Cognition; Non-motor symptoms
MeSH Terms: conditions — Parkinson Disease | interventions — Nordic Walking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dance (Experimental): Dance intervention for 3 months, 2 times/week, 2 hours per week. Dance is a safe and effective form of activity, which has been used in PD population. Participants take part in a dance class specifically for people with PD lead by a qualified dance instructor. The dance class typically include a warm-up, dance related activities developed based on folk and popular dances from the Amazon region in the Brazilian North region and a cool-down.
  Interventions: Behavioral: Amazonian Dance
- Control Group (Active Comparator): Nordic Walking was chosen for the active control group because it is a well accepted, low-cost, safe and effective rehabilitation strategy for PwPD (SALSE-BETÁN et al, 2022).
  Interventions: Behavioral: Nordic Walking

INTERVENTIONS:
Behavioral: Amazonian Dance — Dance intervention consists of 24 Amazonian Dance, 2 times/week, lasting 1 hour, over a period of 12 weeks. Classes will be taught by qualified dance professionals with experience teaching PwPD and will take place in a specific practice room (air-conditioned, spacious, and leveled), with adequate facilities, floors, chairs, bars, mirrors, and sound system.
  Classes will be divided into 4 parts. The part 1 (10-15 min.) consists of welcoming students, warm-up exercises, and body awareness activities. In the Part 2 (10-15 min.) Weight transfer activities, static and dynamic balance, motor coordination, strengthening of lower and upper limbs will be carried out. The part 3 (25-30 min.) will be based on the Amazonian Lundum and Carimbó dances. In the part 4 (5-10 min.), the final part of the class, the calm down activity will be carried out, with breathing, stretching and relaxation activities.
  Arms: Dance
Behavioral: Nordic Walking — The Nordic walking protocol consists of 3 moments: warm-up (10min), main part (40min) and final part (10min). At the beginning of the activity, a joint warm-up is performed and free walking, without poles, at a comfortable speed. Then, in the main part of the class, the participants performed an individual and daily training that is inserted in their general training cycle, elaborated from the specific and individual functional capacity, measured from the application of the 6-minute walk test. In the final part, return to calm and stretching.
  Arms: Control Group

SUMMARY:
This randomized controlled trial aims to evaluate the effects of a 12-week Amazonian dance program on cognitive and motor symptoms in people with Parkinson's disease (PD), comparing outcomes between participants in the intervention and those in an alternative control intervention.

DETAILED DESCRIPTION:
Experimental Design: Randomized controlled single-blind trial with four parallel groups. Study sites include the Federal University of Rio Grande do Sul (South Region, Brazil) and the Federal University of Pará (North Region, Brazil).

Participants: 80 adults aged 50 to 80 years with a clinical diagnosis of idiopathic Parkinson's disease, in stages I-III of the Hoehn & Yahr Scale, under stable pharmacological treatment for at least one year. Participants will be recruited from community health services, Parkinson's associations, and university-affiliated health units in Northern and Southern Brazil.

Interventions:

Amazonian Dance Groups (North and South): Participants will engage in twice-weekly dance sessions for 12 weeks (24 sessions total), including movement practices inspired by Lundum and Carimbó dances, choreographic improvisation, and activities involving memory, storytelling, balance, and mobility.

Control Groups (North and South): Participants will receive a structured non-dance intervention over the same 12-week period. This control activity will consist sessions related to general well-being, physical activity, and quality of life, without dance training.

Outcomes:

Primary Outcome: Cognition (assessed by MoCA, Stroop, and Tab-CAT tools). Secondary Outcomes: Language (TELL), depressive and anxiety symptoms (GDS-15, PAS), quality of life (PDQ-39), functional mobility (TUG), fear of falling (FES-I), and freezing of gait (FOGQ). Experience with Dance, Sociodemographic and clinical data will also be collected.

Data Analysis: Descriptive statistics will report means and standard deviations. Group comparisons over time will be analyzed using Generalized Estimating Equations (GEE) with Bonferroni post-hoc tests. Statistical significance is set at p<0.05. Effect sizes will be interpreted using Cohen's d (small = 0.2, medium = 0.5, large = 0.8), with 95% confidence intervals reported. Analyses will include intention-to-treat, considering participants with at least 80% adherence.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PD according to the London Brain Bank Criteria;
* Able to understand the verbal instructions for the tests;
* Hoehn and Yahr (H&Y) stages I-III
* ≥ 1 year undergoing medical treatment for PD with regular use of anti-parkinsonian drugs
* Capability to participate will be based on the Unified Parkinson's Disease Rating Scale -motor examination

Exclusion Criteria:

* Recent surgeries,
* Deep brain stimulation (DBS);
* Other associated neurological diseases or chronic diseases
* Fitted with a pacemaker;
* Prostheses in the lower limbs;

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2025-11-26 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognition | Change from baseline at 3 months
  Cognition will be assessed in two ways using traditional pen-and-paper tests and incorporating innovative instruments and using digital technology. Executive function and attention will be measured using the Tablet-based Cognitive Assessment (Tab-CAT) application, developed for the efficient detection of mild neurocognitive disorders, which assesses cognitive abilities including memory, executive/speed, visuospatial and language (Possin et al., 2018). In this battery, the Dot-counting, Set-shifting, Flanker, and Animal Fluency tests will be used. The Montreal Cognitive Assessment (MoCA) Brazilian version (Hobson, 2015) will be used to screen for mild cognitive impairment, accessing different cognitive domains in the following areas: attention and concentration, executive functions, memory, language, visuoconstructive skills, conceptualization, calculation and guidance. The total MoCA score is 30 points, with a score of 26 or more considered normal.
1.1 - Cognition - Dot-couting | Change from baseline at 3 months
  This task assesses sustained attention and working memory. The participant is presented with various screens containing different sets of shapes and is instructed to count a specific type. In addition to counting, the participant must remember the totals across multiple trials, which requires continuous focus and short-term retention. This task is sensitive to impairments in attentional and memory systems, often affected in neurological conditions.
1.2 - Cognition - Set-shifting | Change from baseline at 3 months
  This task aims to assess executive shifting, one of the cognitive functions involved in mental flexibility. The stimuli consist of geometric shapes (rectangle or triangle) in different colors (red or blue). During the test, the participant sees a cue word displayed in the center of the screen-either "color" or "shape". Above this cue, a target stimulus (a colored shape) appears. In the lower left and right corners of the screen, two response options are shown, each representing a different combination of shape and color. The participant must select the correct option based on the instruction word shown-i.e., they must match the target either by color or by shape, alternating between these classification rules depending on the cue presented on each trial.
1.3 - Cognition - Flanker | Change from baseline at 3 months
  The Flanker Task is used to assess selective attention and inhibitory control. The participant sees a row of five arrows and must quickly indicate the direction of the central arrow (the target), while ignoring the surrounding arrows (flankers). These flankers may be congruent (pointing in the same direction) or incongruent (pointing in the opposite direction). The task measures the individual's ability to suppress irrelevant stimuli and respond accurately to the target, making it a valuable tool for detecting deficits in executive control.
1.4 - Cognition - Animal Fluency | Change from baseline at 3 months
  In this task, the participant is asked to name as many animals as possible in one minute. It evaluates semantic verbal fluency and is highly sensitive to early dysfunction in brain regions associated with language, particularly in the frontotemporal areas.
1.5 - Cognition - MoCA | Change from baseline at 3 months
  The MoCA (Montreal Cognitive Assessment) was used to assess global cognition. In Brazil, the interpretation of MoCA scores varies according to educational level and group differences (Cesar et al., 2019). The MoCA cutoff score to differentiate cognitively unimpaired (CU) from people with dementia is 15. To distinguish cognitively unimpaired (CU) from people mild cognitive impairment (MCI), the cutoff score is 19. Furthermore, the MoCA cutoff score for identifying MCI varies according to individuals' educational levels, reflecting the importance of tailoring assessments to educational contexts. For individuals with no formal education, the cutoff score is 11.5. Those with 1 to 4 years of education have a cutoff score of 18. Individuals with 5 to 8 years of education have a cutoff score of 19.5, as do those with 9 to 11 years of schooling. Finally, for individuals with 12 or more years of education, the cutoff score is 22. These values underscore the need to consider educational context
Language | Change from baseline at 3 months
  The Toolkit to Examine Lifelike Language (TELL) will be used in this study to assess elements of language and speech. This application enables the recording, storage, and encryption of participants' oral productions. Speech samples will be recorded in Wave format (.wav) with an optimal sampling rate of 44.1 kHz and bit depth of 24 bits. Transcriptions will be performed automatically via Whisper, integrated within the TELL platform, and manually reviewed according to standard criteria established in previous studies (Steeb et al., 2018). Both audio files and transcriptions will undergo pre-processing using validated pipelines, allowing for the extraction of linguistic and acoustic features. These automated methods will be employed to identify distinct speech patterns, as described by Garcia et al. (2022). In addition, the tools used in the study offer potential to assess and monitor disease progression and treatment effectiveness in relation to verbal communication (Garcia et al, 2016)

SECONDARY OUTCOMES:
Anxiety symptoms | Change from baseline at 3 months
  Anxiety disorders will be assessed using the Parkinson Anxiety Scale (PAS), an instrument specifically developed to assess anxiety in PwPD (Leentjens et al., 2014). This scale consists of 12 questions, each of which can be scored from zero (0) to four (4), totalling a maximum score of 48 points. It is divided into the persistent anxiety subscale (AF; 1st to 5th questions), which measures generalized anxiety disorders; the episodic anxiety subscale (EA; 6th to 9th questions), which assesses panic disorder; and the avoidance behaviour subscale (AB; 10th to 12th questions), which assesses anxious symptoms of agoraphobia and social phobia.
Depressive symptoms | Change from baseline at 3 months
  For the evaluation of depressive symptoms, the Geriatric Depressive Symptoms (GDS-15) will be used, which is a scale widely used and validated as a diagnostic tool for depression in the elderly, classified into mild, moderate and severe levels. It is a scale for assessing depressive symptoms, self-assessed, consisting of 15 questions, in which the result of five or more points is indicative of a probable depressive episode. (Paradela et al., 2005).
Quality of life symptoms | Change from baseline at 3 months
  Quality of life will be measured by applying the Parkinson's Disease Questionnaire - 39 (PDQ-39), proposed and validated by Peto et al. (1995). The PDQ-39 comprises eight domains: mobility, daily life activities, emotional well- being, stigma, social support, cognition, communication, and bodily discomfort. Each item can be answered according to five predetermined answers: never; rarely; sometimes; often; always. The score of each item ranges from 0 to 4 points, and the total score varies from 0 to 100 points, where the lowest scores reflect a higher quality of life (Marinus et al., 2002; Lana et al., 2007).
Levels of Hope | Change from baseline at 3 months
  To assess the levels of hope, the Herth Hope Scale will be used, which has 12 affirmatively written items where the items are graded on a 4-point Likert-type scale, ranging from completely agree to completely disagree, where 1 indicates completely disagree and 4 indicates completely agree. The total score ranges from 12 to 48 and the higher the score, the higher the level of hope (Sartore & Grossi, 2008).
Functional Mobility | Change from baseline at 3 months
  In the Timed up and Go (TUG) test, participants will start sitting in a chair with their arms crossed over their chest, knees, hips and feet at a 90º angle, with their feet placed parallel, and instructed to stand up, uncross their arms, walk a distance of 3 meters, pass in a cone (180º turn), go back and sit on the chair crossing your arms over your chest (Podsiadlo & Richardson, 1991). Participants will perform the TUG test three times, at two speeds (SSS and FS). The best result of the three repetitions at each speed will be considered.
Fall symptoms | Change from baseline at 3 months
  The Falls Efficacy Scale - International (FES-I) works as an indicator of the possible occurrence of a fall event and is composed of 16 items that establish the risk of falling for each elderly person within their life context, during basic daily life activities and instrumental/social, on a four-point scale. The total score varies between 16 points (not worried) and 64 points (very worried). (Yardley et al., 2005).
Gait freezing | Change from baseline at 3 months
  The Freezing of Gait Questionnaire (FOGQ) consists of six questions about gait freezing episodes: duration, frequency of freezing, hesitation, walking in the worst state of walking, and whether these events affect functional independence and activities of daily living. It has a total score of 24, with the highest score representing severe gait impairment (Baggio et al., 2012).

OTHER OUTCOMES:
PD motor symptoms | Change from baseline at 3 months
  Part III of the MDS-UPDRS (Movement Disorder Society - Unified Parkinson's Disease Rating Scale) will be used in this study to assess participants' motor impairment. This section includes 18 items that evaluate speech, facial expression, resting and postural tremors, rigidity, hand and leg agility, posture, gait, balance, and dyskinesias. Each item is scored from 0 to 4, with a total score ranging from 0 (normal function) to 56 (greater motor impairment) (Goetz et al., 2021; Mello & Botelho, 2010).
Experience with Dance | baseline
  The Goldsmith's Dance Sophistication Index (Gold-DSI) is used to assess the participants' level of dance experience. Twenty items assess experience in dance participation along four subscales: body awareness (six items), social dancing (six items), urge to dance (five items), and dance training (three items). The general factor dance participation comprises all 20 items from the four subscales. The mean of range values (i.e., 1 to 7) reflects the result of each subscale or general factor, with higher scores (i.e., those near to 7) indicating higher dance sophistication. A further six items measure experience in watching dance. This questionnaire provides a brief, standardized, and continuous evaluation of doing, watching, and knowing about dance (Rose, Müllensiefen, Lovatt & Orgs, 2022).

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Universidade Federal do Pará, Castanhal, Pennsylvania
  - Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No